CLINICAL TRIAL: NCT06222463
Title: Power Dissipation in Low Tidal Volume Versus Individualized Flow-controlled Ventilation - a Randomized, Clinical Cross-over Trial
Brief Title: Power Dissipation in Flow-controlled Ventilation
Acronym: POWER-FLOW
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1091/2023
Record Dates: First submitted 2024-01-16; First posted 2024-01-24 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-01

CONDITIONS: Mechanical Ventilation; Abdominal Surgery
Keywords: Flow-controlled Ventilation; Power Dissipation; Mechanical Power

STUDY DESIGN:
Intervention Model Description: non-blinded, randomized, cross-over, controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low tidal volume ventilation (Active Comparator): Flow-controlled ventilation will be established with a PEEP of 5 cmH2O, peak pressure set to achieve a tidal volume of 7 ml/kg predicted body weight and the flow set to achieve normocapnia at an I:E ration of 1:1. Three consecutive measurements of power dissipation with 15 minutes in between will be obtained. Additionally secondary outcome parameters such as respiratory parameters and results of arterial blood gas analysis will be recorded at each measurement timepoint.
  Interventions: Device: Evone
- individualized FCV (Experimental): Flow-controlled ventilation will be individualized with compliance guided PEEP and peak pressure titration. The flow will be set to achieve normocapnia at an I:E ration of 1:1. Three consecutive measurements of power dissipation with 15 minutes in between will be obtained. Additionally secondary outcome parameters such as respiratory parameters and results of arterial blood gas analysis will be recorded at each measurement timepoint.
  Interventions: Device: Evone

INTERVENTIONS:
Device: Evone — Evone (Ventinova Medical B.V., Eindhoven, The Netherlands) is a ventilator, which is able to perform flow-controlled ventilation (FCV). Moreover it provides direct tracheal pressure measurements and combined with the constant gas flow of FCV a precise determination of dynamic compliance is feasible. Thus not only PEEP but also peak pressure can be titrated based on dynamic compliance. Additionally intratracheal pressure-volume loops can be measured and thus power dissipation calculated, which represents the primary outcome parameter of this trial.

SUMMARY:
The goal of this randomized clinical cross-over trial is to compare power dissipation (Pd) during flow-controlled ventilation with either standard of low tidal volume ventilation or compliance guided individualization of ventilator settings. This study is performed in patients scheduled for open abdominal surgery and the primary and secondary outcome parameters are:

* power dissipation [J/min] during ventilation calculated by integrating the hysteresis of the tracheal pressure-volume loop
* applied mechanical power during ventilation calculated by published formulas [1]
* oxygenation of the blood assessed by PaO2/FiO2 ratio
* decarboxylation assessed by required respiratory minute volume to maintain normocapnia
* comparison of respiratory variables in low tidal volume versus individualized ventilation Participants will randomly receive either low tidal volume (LTV) or individualized flow-controlled ventilation [2]. In the LTV group, the positive end-expiratory pressure will be set to 5 cmH2O and the peak pressure set to achieve a tidal volume of 7 ml/kg predicted body weight. In the individualized group positive end-expiratory and peak pressure will be titrated to achieve the highest compliance [2]. In both groups the flow will be set to achieve normocapnia (PaCO2 35-45 mmHg). After obtaining three consecutive measurements the ventilation strategy will be switched to the alternative regime in a cross-over design and again, three measurements recorded.

The investigators hypothesize, that individualized ventilator settings are able to improve ventilation efficiency in terms of a lower required minute volume to maintain normocapnia and thus is able to reduce power dissipation during ventilation. Secondary endpoint will be a comparison of Pd to calculated mechanical power, as a currently accepted surrogate parameter for ventilation invasiveness [2] and also outcome predictor. Additionally, gas exchange parameters such as oxygenation and decarboxylation will be compared between low tidal volume and individualized ventilation.

DETAILED DESCRIPTION:
After anesthesia induction and securing the airway with a tracheal tube, tha patients will be ventilated with flow-controlled ventilation (FCV) using standard of low tidal volume ventilation with a positive end-expiratory pressure (PEEP) of 5 cmH2O and the peak pressure set to achieve a tidal volume of 7 ml/kg predicted body weight. I:E ration will be set to 1:1, the gas flow adjusted to achieve normocapnia and the fraction of inspired oxygen adjusted to achieve normoxia. After opening the abdominal cavity baseline parameters will be recorded and subsequently the study participant randomized to one of the following treatment group:

* low tidal volume ventilation (LTV): PEEP will be set to 5 cmH2O, peak pressure adjusted to achieve a tidal volume of 7 ml/kg predicted body weight and the flow set to achieve normocapnia (PaCO2 of 35-45 mmHg)
* individualized FCV: PEEP and peak pressure will be titrated based on dynamic compliance. First PEEP well be increased or decreased until the highest tidal volume at the same driving pressure can be achieved. Then the driving pressure or peak pressure will be increased, until there is no further over-proportional increase in tidal volume (previous tidal volume + measured compliance). Finally the gas flow will be set to achieve normocapnia (PaCO2 of 35-45 mmHg) Three measurements will be obtained with 15 minutes in between and subsequently the ventilation setting switched to the alternative group, followed by additional three consecutive measurements. After obtaining all study related measurements the observation period ends and the patient will be further treated with the ventilation strategy that results in the lowest energy dissipation.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects ≥ 18 years
* Body weight ≥ 40 kg
* Elective open abdominal surgery under general anaesthesia - American Society of Anesthesiologists Classification I-III
* Written informed consent

Exclusion Criteria:

* Emergency surgery
* American Society of Anesthesiologists Classification IV-V
* Female subjects known to be pregnant
* Known participation in another interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Power dissipation (Pd) | Pd will be calculated and recorded three times in each treatment arm with 15 minutes in between.
  The hysteresis of the tracheal pressure-volume relationship represents the power, that is dissipated during one ventilation cycle. Together with the respiratory rate, overall power dissipation can be calculated in J/min.

SECONDARY OUTCOMES:
Mechanical power (MP) | MP will be calculated and recorded three times in each treatment arm with 15 minutes in between.
  Applied mechanical power during inspiration will be calculated based on a published formula by Gattinoni et al.
PaO2/FiO2 ratio | PaO2/FiO2 ratio will be measured and recorded three times in each treatment arm with 15 minutes in between.
  Oxygenation will be assessed with the help of an arterial blood gas analysis
Minute volume (MV) | MV will be recorded three times in each treatment arm with 15 minutes in between
  Required respiratory minute volume to maintain normocapnia will be recorded.

OTHER OUTCOMES:
Respiratory measurement variables | Respiratory measurement variables will be recorded three times in each treatment arm with 15 minutes in between
  Ventilator settings and readings with positive end-expiratory pressure, peak pressure, respiratory rat, flow rate, compliance and resistance will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Spraider, PhD, Principal Investigator — Medical University of Innsbruck, Department of Anesthesia and Intensive Care Medicine
Locations (1):
- Medical University of Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No
The IPD can be requested from the principal investigator.

REFERENCES:
- [Background] Gattinoni L, Tonetti T, Cressoni M, Cadringher P, Herrmann P, Moerer O, Protti A, Gotti M, Chiurazzi C, Carlesso E, Chiumello D, Quintel M. Ventilator-related causes of lung injury: the mechanical power. Intensive Care Med. 2016 Oct;42(10):1567-1575. doi: 10.1007/s00134-016-4505-2. Epub 2016 Sep 12. PMID 27620287
- [Background] Spraider P, Abram J, Martini J, Putzer G, Glodny B, Hell T, Barnes T, Enk D. Flow-controlled versus pressure-controlled ventilation in cardiac surgery with cardiopulmonary bypass - A single-center, prospective, randomized, controlled trial. J Clin Anesth. 2023 Dec;91:111279. doi: 10.1016/j.jclinane.2023.111279. Epub 2023 Oct 3. PMID 37797394